CLINICAL TRIAL: NCT05858164
Title: An Open-label, Phase 1, First-in-human, Dose Escalation Study to Evaluate the Safety, Tolerability, Maximum Tolerated or Administered Dose, Pharmacokinetics, Pharmacodynamics, and Tumor Response Profile of the Diacylglycerol Kinase Alpha Inhibitor (DGKαi) BAY 2862789 in Participants With Advanced Solid Tumors
Brief Title: A First-in-human Study to Learn How Safe the Study Treatment BAY2862789 is, to Find the Best Dose, How it Affects the Body, What Maximum Amount Can be Given, How it Moves Into, Through and Out of the Body, and How it Acts on Different Tumors in Participants With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 22231; 2024-510998-26-00 (Other: CTIS (EU))
Record Dates: First submitted 2023-05-05; First posted 2023-05-15 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Advanced Solid Tumors; Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Dose Escalation (Experimental): Participants will take BAY2862789 oral doses.
  Interventions: Drug: BAY2862789

INTERVENTIONS:
Drug: BAY2862789 — Oral administration, solution or tablets

SUMMARY:
Researchers are looking for a better way to treat people who have advanced solid tumors including a specific kind of lung cancer (non-small cell lung cancer, NSCLC).

Advanced solid tumors are types of cancer that have spread to nearby tissue, lymph nodes, and/or to distant parts of the body and that are unlikely to be cured or controlled with currently available treatments.

BAY2862789 works by blocking an enzyme in T-cells, thereby activating them. T-cells are a type of immune cell that are known to have an anti-cancer effect.

The main purpose of this first-in-human study is to learn:

* how safe different doses of BAY2862789 are,
* the degree to which medical problems caused by BAY2862789 can be tolerated (also called tolerability),
* what maximum amount (dose) can be given, and
* how BAY2862789 moves into, through and out of the body.

To answer this, the researchers will look at:

* the number and severity of medical problems participants have after taking BAY2862789 for each dose level. These medical problems are also referred to as adverse events. An adverse event is considered "serious" when it leads to death, puts the participants' lives at risk, requires hospitalization, causes disability, causes a baby being born with medical problems or is otherwise medically important.
* the (average) total level of BAY2862789 in the blood (also called AUC) after intake of single and multiple doses.
* the (average) highest level of BAY2862789 in the blood (also called Cmax) after intake of single and multiple doses.

Doctors and their team keep track of all medical problems that participants have during the study, even if they do not think the medical problem might be related to the study treatment.

In addition, the researchers want to know if and how the participants' tumors change after taking BAY2862789.

The dose escalation will be done to find the most appropriate dose that can be given. For this, each participant will receive one of the increasing doses of Bay 2862789. More groups might be investigated based on new data that emerges. For this, each participant will receive one of the increasing doses of BAY2862789.

Participants in the study will take the study treatment until their tumor gets worse (also known as 'disease progression'), until they have medical problems, until they leave the study, or until the study is terminated.

Each participant will be in the study for several months, including a test (screening) phase of up to 28 days, few months of treatment depending on the participant's benefit, and a follow up phase after the end of treatment. The following approximate numbers of visits to the study site are planned: two during the screening phase, six in the first treatment month, one to three per month in the following periods.

During the study, the study team will:

* take blood and urine samples
* do physical examinations
* check vital signs such as blood pressure, heart rate, body temperature
* examine heart health using ECG (electrocardiogram)
* check cancer status using CT (computed tomography) or MRI (magnetic resonance imaging) and, if needed, bone scans
* take tumor samples (if required)
* pregnancy test

The treatment period ends with a visit no later than 7 days after the last BAY2862789 dose. The study doctors and their team will check the participants' health and any changes in cancer about 30 and 90 days after the last dose and every 12 weeks thereafter. This follow-up period ends if the cancer worsens, if a new anti-cancer treatment is started, or until the participant leaves the study. In addition, the study doctors and their team will contact the participant every 12 weeks to learn about the participant's survival. This ends no later than 12 months after the last participant started treatment or by the end of the study, whichever comes first.

If the study participant benefits from treatment, continuation of treatment with BAY2862789 beyond the duration of this study might be possible.

ELIGIBILITY:
Inclusion Criteria:

* Capable of giving signed informed consent
* Be ≥18 years of age on day of signing informed consent.
* Have measurable disease per Response Evaluation Criteria in Solid Tumours version 1.1 (RECIST 1.1) as assessed by the local site investigator.
* Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1.
* Participants with a histologically confirmed diagnosis of a solid tumor that have exhausted available treatments known to be beneficial for this tumor type or for whom these treatments are not acceptable and for whom this trial is a reasonable option for them, will be enrolled onto this study. Appropriate molecular profiling of tumors should have been performed according to local national guidelines prior to trial entry. Specifications for the different parts of the study are below:

  -- Dose escalation: All solid cancers, except primary central nervous system cancers.
* Provision of archival tumor sample at baseline is mandatory for all participants in escalation, and expansion cohorts.
* Participants must be willing to undergo mandatory paired biopsies of tumor (pre- and on- treatment).
* Have adequate organ function.
* Agree to use contraception during the treatment period and for at least 6 months after the last dose of study treatment.

Exclusion Criteria:

* Had an allogeneic tissue/solid organ transplant.
* Previous therapy with a diacylglycerol kinase (DGK) inhibitor
* Has received a prior therapeutic regimen containing an anti-programmed cell death protein 1 (anti-PD-1), anti-programmed death-ligand 1 (anti-PD-L1), or anti-programmed cell death 1 ligand 2 (anti PD-L2) agent or an agent directed to another stimulatory or co-inhibitory T-cell receptor (e.g., cytotoxic T-lymphocyte-associated protein 4 (CTLA-4), OX 40, CD137) and was discontinued from that treatment regimen due to a Grade 3 or higher immune related adverse event (irAE) or any toxicity that was life-threatening.
* Has received prior systemic anti-cancer therapy including investigational agents within 4 weeks or 5 half-lives, whatever is shorter, prior to treatment. Growth factor treatments such as granulocyte colony-stimulating factor (G-CSF) must have been discontinued 4 weeks prior to entering the study.
* Participants must have recovered from previous radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis.
* Participants cannot have had a blood transfusion within 2 weeks of starting therapy.
* Has received a live vaccine within 30 days prior to the first dose of study drug.
* Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study treatment.
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug.
* Has a known additional malignancy that is progressing or has required active treatment within the past 3 years.
* Participants with new brain metastases on screening brain magnetic resonance imaging/computed tomography (MRI/CT).
* Primary central nervous system malignancy or presence of leptomeningeal disease.
* Participants with gastrointestinal conditions that may compromise oral absorption such as short bowel syndrome or active tumor-related bowel obstruction with ongoing symptoms compromising absorption over last 6 months.
* Has an active autoimmune disease including inflammatory bowel disease that has required systemic treatment in past 2 years.
* Current pneumonitis / interstitial lung disease.
* Has an active infection requiring systemic therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2023-08-07 (Actual); Primary Completion 2025-09-26 (Actual); Study Completion 2025-09-26 (Actual)

PRIMARY OUTCOMES:
The number and severity of treatment-emergent adverse events (TEAEs) | Up to 90 days after the last administration of the study treatment
  Adverse events (AEs) will be considered treatment-emergent if they have started or worsened after first administration of study treatment up to 90 days after the last administration of study treatment.
Number of participants experiencing dose-limiting toxicities (DLTs) at each dose level in the Dose Escalation part of the study | Up to 21 days after the first administration of the study treatment
Recommended Dose for Expansion (RDE) | Up to 2 years
  RDE: as determined by safety, tolerability, pharmacokinetics (PK), and pharmacodynamics (PD) and efficacy data
Maximum concentration (Cmax) BAY2862789 after single-dose | from pre-dose up to 24 hours after administration on Cycle 1 Day 1 (each cycle is 21 days)
Maximum concentration (Cmax) BAY2862789 after multiple-dose | Pre-dose and up to 24 hours after Day 16 in Cycle 1
Area under the curve (AUC) BAY2862789 after single-dose | from pre-dose up to 24 hours after administration on Cycle 1 Day 1 (each cycle is 21 days)
Area under the curve (AUC) BAY2862789 after multiple-dose | Pre-dose and up to 24 hours after Day 16 in Cycle 1

SECONDARY OUTCOMES:
Objective response rate (ORR) | Up to 2 years
  ORR is defined as the proportion of participants whose best overall response is either a confirmed complete response (CR) or confirmed partial response (PR) according to Response Evaluation Criteria in Solid Tumours version 1.1 (RECIST 1.1) (investigator assessed).
Disease control rate (DCR) | Up to 2 years
  DCR is defined as the percentage of participants whose best overall response was either CR, PR, or SD, considering the requirement for confirmation of CR and PR.
  CR stands for complete response. PR stands for partial response. SD stands for stable disease.
Duration of response (DOR) | Up to 2 years
  DOR is defined as the time from the first documented objective response of PR or CR, whichever occurs earlier, to disease progression or death (if death occurs before progression is documented).
  PR stands for partial response. CR stands for complete response.
Progression-free survival (PFS) at 6 months | Up to 6 months
  PFS is defined as the time from the start of study treatment to the date of first observed disease progression by investigator assessment or death due to any cause, if death occurs before progression is documented.
Overall survival (OS) at 12 months | Up to 12 months
  OS is defined as the time from the start of study treatment to death due to any cause.
Activation of effector T memory cells | Up to 2 years
Ex vivo stimulated short-term activation of Interleukin 2 (IL2) and interferon-gamma | Up to 2 years

CONTACTS AND LOCATIONS:
Locations (18):
- United States (5):
  - AdventHealth medical Group Oncology Research at Celebration, Celebration, Florida
  - Brigette Harris Cancer Pavilion at Henry Ford Cancer Center - Detroit, Detroit, Michigan
  - Cancer Center and Research Institute - UMMC, Jackson, Mississippi
  - The University of Texas MD Anderson Cancer Center - Texas Medical Center, Houston, Texas
  - START | San Antonio, San Antonio, Texas
- Australia (2):
  - The Kinghorn Cancer Centre - Medical Oncology Department, Darlinghurst, New South Wales
  - Princess Alexandra Hospital Australia, QLD, Queensland
- China (2):
  - Tongji Hosp. of Tongji Med Coll, Huazhong Uni of Sci & Tech., Wuhan, Hubei
  - Jilin Cancer Hospital, Changchun, Jilin
- Israel (2):
  - Hadassah Hebrew University Hospital Ein Kerem, Jerusalem
  - Tel-Aviv Sourasky Medical Center, Tel Aviv
- South Korea (5):
  - Gyeongsang National University Hospital, Jinju, Gyeongsangnam-do
  - Chungbuk National University Hospital, Cheongju-si, North Chungcheong
  - Asan Medical Center - Oncology Department, Seoul, Seoul Teugbyeolsi
  - Seoul National University Hospital, Seoul, Seoul Teugbyeolsi
  - The Catholic University of Korea Seoul St. Mary's Hospital, Seoul
- Spain (2):
  - Hospital Universitari Vall d'Hebron - Institut d'Oncologia - Grupo de Tumores Toracicos y Cancer de Cabeza y Cuello, Barcelona
  - Hospital Universitario Virgen De La Victoria - Oncology, Málaga

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.

REFERENCES:
- See also: Click here to find information for studies related to Bayer products. To find this study enter the ClinicalTrials.gov identifier (NCT) number or Bayer Study Identifier (ID) in the search field. — https://clinicaltrials.bayer.com/study/22231/